CLINICAL TRIAL: NCT01948531
Title: Clinical and Instrumental Evaluation of a Topical "Antiage" Formulation for the Face
Brief Title: Clinical Trial on a Topical "Antiage" Face Gel
Acronym: E2912
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DermIng E2912
Record Dates: First submitted 2012-12-10; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Wrinkles
Keywords: Antiage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gynomunal® gel (Experimental): The study will be conducted on 33 healthy volunteers of female sex aged between 35 and 65 years old; each subject will apply a fixed quantity of the Gynomunal gel on the face (including the submental area) twice a day, in the morning and in the evening (preferentially always at the same hour), with a mild massage.
  Interventions: Drug: Gynomunal® gel

INTERVENTIONS:
Drug: Gynomunal® gel — A fixed quantity of the cosmetic product will be applied on the face (including the submental area) twice a day, in the morning and in the evening (preferentially always at the same hour), with a mild massage according to the instructions received by the investigator during the basal visit (T0).
  Other Names: Ialuronic acid gel

SUMMARY:
Aim of the study is to evaluate clinically and by non-invasive instrumental evaluations the "antiage" activity of Gynomunal® gel after one single application on the face (short term evaluation) and 4 weeks of repeated use twice daily (long term evaluation) by healthy female volunteers.

It is also aim of this study to evaluate cosmetic acceptability by the volunteers and efficacy and tolerance both by investigator and volunteers.

DETAILED DESCRIPTION:
Controlled clinical trial that foresees the application of the study product for an uninterrupted period of 4 weeks. 4 visits will be performed: a basal visit (T0), a short term evaluation 20 minutes after the 1st product application (T20min) and a long term evaluation after 2 (T2 - intermediate visit) and 4 (T4 - final visit) week-treatment.

The study will be conducted on 33 healthy volunteers of female sex, 11 women for each of the following groups:

* 35-44 years
* 45-54 years
* 55-65 years The volunteers accept to respect the rules fixed in the list of recruitment criteria and not to deviate from their normal life habits. Moreover, the month preceding the inclusion visit and during the entire period of treatment, normal cleansing habits must be maintained, sun and UV light exposure, avoided. In the case of UV exposure must be used a sun screen total block cream.

Each volunteer is precisely informed about the study, a consent form being completed and signed. At the end of the study the investigator will declare to have informed all the volunteers participating it, signing and dating the relative form.

The study will be started only after Independent Ethical Committee approval. It is understood that the treatment would be immediately interrupted as soon as the investigator judges it necessary.

For each volunteer a Case Record Form is filled and to each one a progressive number is assigned. Personal data, subject's history, clinical and instrumental evaluations are registered in basal conditions and at all study visits.

During 3 hours before the visit the volunteer must not smoke, drink coffee or alcohol. Any cosmetic product can be used on the skin test area during 2 hours before the visit. All measurements are performed under standard environmental conditions (Temperature=22+\-2°C; Relative Humidity<60%).

Before each visit the volunteer will get acclimatized under relax conditions for at least 10-15 min.

Each volunteer will report on the personal diary card all information about the date, the time of study product application and a comment if necessary.

At each visit, the volunteers must give back the diary card to the Investigator to verify their compliance.

Samples are handled by DermIng in accordance with the methods described in the company operating procedures (SOP).

This trial is carried out by DermIng in accordance with the methods described in its own company operating procedures (SOPs). The information and data on the trial are generated, recorded, documented and processed in accordance with the methods described in the following procedure, based on ICH GCP 1996. The trial is covered by an insurance policy provided by Polichem S.A. to cover any damages related to the study product.

Statistical plan: the activity of the test product at T20min, T2 and T4 will be expressed in absolute values versus baseline (T0) for the entire population and for each evaluated group (35-44 yeas, 45-54 years, 55-65 years). Moreover a comparison between groups will be carried out at each considered time. Clinical data The statistical analysis of clinical data is carried out with not parametric test, while the analysis of all instrumental data are carried out with parametric test.

ELIGIBILITY:
Inclusion Criteria:

* female healthy subjects;
* age 35-65 years;
* presence of light-moderate face ritidosis;
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, face cleansing and make- up use;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study;
* accepting to sign the Informed consent form

Exclusion Criteria:

* Pregnancy;
* lactation;
* change in the normal habits regarding foods, physical activity, face cleansing and make-up use during the month preceding the test;
* sensitivity to the test product or its ingredients;
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study actually or during the previous 3 months;
* change in the normal life habits during the month preceding the inclusion.
* dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Wrinkles profilometry (Ra - micrometers) | 4 weeks
  A picture of crow's feet area is taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to elaborate 3D representations of skin wrinkles as well as to measure skin principal profilometric parameters in vivo or on skin replicas.
  As a measuring method Primos compact uses a digital stripe projection based on micro mirrors which allows for fast and highly precise measuring data acquisition (the speed of under 70ms for the measuring data admission provide perfect results of measurement).

SECONDARY OUTCOMES:
Plastoelasticity | 4 weeks
  Among the various methods studied in order to measure the skin elasticity grade, the torsion one is the most effective, as it is very sensible to the variations of the mechanical properties of the corneum stratum. Skin firmness is measured with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK). This instrument is based on the principle of the torsion given to the skin surface by a probe made of two circles that adhere to the skin through shaped adhesive tapes. The internal circle rotation, while the external circle is still, exerts a constant torsion of the skin (torsion time = 1 second with a torque = 9mN*m). The instrument measures the torsion angle (θ) during the mechanical stimulus ("torque on") and after it has ceased ("torque off").
  Parameters:
  Ue: immediate extensibility ("torque on" at 0.02 sec.) Uf: maximum extensibility ("torque on" at 0.9 sec.) Uv: viscoelasticity Ur: immediate elastic recovery ("torque off" at 0.02 sec.).
Electrical capacitance of skin (hydration) | 4 weeks
  Hydration is measured by the instrument Corneometer CM825 (Courage - Khazaka, Köln, Germany): a square sensor (49mm2) frontally covered by a special glass, mounted on a spring cursor able to measure electrical capacity. Leaning the sensor on the skin surface, with a constant pressure thanks to the spring cursor it is possible to perform measures. The sensor acts as a capacitor. When a voltage is applied to this capacitor, the quantity of electric charge stored will be dependent on the dielectric properties of the material in contact with the probe. Water has an unusually high dielectric constant and so its presence in the skin is readily detectable by this method. So the measure of the skin capacitance properties is an indirect expression of its hydration level.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Medical Doc, Principal Investigator — Derming SRL
Locations (1):
- DermIng S.r.l. Single Member Company, Monza, MB, Italy